CLINICAL TRIAL: NCT04107298
Title: A Prospective, Multi-Center, Single-Arm, Feasibility Study to Assess the Safety and Performance WIth the SUNDANCE™ DruG Coated Balloon for the Treatment of De Novo or Restenotic Lesions in Infra-Popliteal Arteries
Brief Title: Safety and Feasibility of Surmodics SUNDANCE™ Drug Coated Balloon
Acronym: SWING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SurModics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUR19-002
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease; Critical Lower Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- SUNDANCE™ Drug Coated Balloon (Experimental): SUNDANCE™ Drug Coated Balloon
  Interventions: Device: SUNDANCE™ Drug Coated Balloon

INTERVENTIONS:
Device: SUNDANCE™ Drug Coated Balloon — Angioplasty procedure with a sirolimus-coated, percutaneous transluminal angioplasty (PTA) balloon catheter

SUMMARY:
To evaluate the safety and performance of the Sundance™ DCB in subjects with occlusive disease of the infrapopliteal arteries.

DETAILED DESCRIPTION:
SWING is a prospective, multi-center, single-arm, feasibility study to assess the safety and performance of the Sundance™ drug coated balloon for the treatment of de novo or restenotic lesions in infra-popliteal Arteries. Approximately 35 subjects will be treated at up to 8 sites.

ELIGIBILITY:
Clinical Inclusion Criteria

* Subject is ≥18 years.
* Subject has target limb Rutherford classification 4 or 5. Rutherford classification 3 subjects may be enrolled but will be capped to a limit of 20% of the total enrollment (i.e., no more than 7 Rutherford class 3 subjects may be enrolled in the study).
* Subject has provided written informed consent and is willing to comply with study follow-up requirements.

Clinical Exclusion Criteria

* Subject has acute limb ischemia.
* Subject underwent intervention involving the target vessel (not a proximal inflow vessel) within the previous 90 days.
* Subject previously underwent PTA of the target lesion vessel using a DCB or DES.
* Subject has had prior vascular intervention in the contralateral limb within 14 days before the planned study index procedure or subject has planned vascular intervention in the contralateral limb within 30 days after the index procedure.
* Subjects with heel gangrene, deep heel ulcers, osteomyelitis of tarsal or metatarsal bones (which extends beyond the metatarsal head immediately adjacent to the metatarso-phalangeal joint), and subjects with exposed vital structures (e.g., medial or lateral malleolus).
* Subjects requiring pedal angioplasty.
* Subjects that are non-ambulatory and confined to bed.
* Women who are pregnant, breast-feeding or intend to become pregnant or men who intend to father children during the time of the study.
* Subject has history of Class 3 (and above) congestive heart failure (CHF) in past 6 months.
* Subject has life expectancy less than 12 months.
* Subject has a known allergy to contrast medium that cannot be adequately pre-medicated.
* Subject has known hypersensitivity to sirolimus
* Subject has a known contraindication to the intended concomitant medications.
* Subject is allergic to ALL antiplatelet treatments.
* Subject has impaired renal function (i.e. serum creatinine level ≥2.5 mg/dL or ≥221 µmol/L).
* Subject had major limb amputation on the affected side in last year or has planned major limb amputation.
* Subject is receiving immunosuppressant therapy.
* Subject has known or suspected active infection at the time of the index procedure.
* Subject has platelet count <100,000/mm3 or >700,000/mm3.
* Subject has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the study procedure.
* Subject is diagnosed with coagulopathy or other disorders which are contraindications for treatment with systemic anticoagulation and/or dual antiplatelet therapy (DAPT).
* Subject has history of stroke within the past 3 months.
* Subject has a history of myocardial infarction within the past 30 days.
* Subject is unable to tolerate blood transfusions because of religious beliefs or other reasons.
* Subject is incarcerated, mentally incompetent, or abusing drugs or alcohol.
* Subject is participating in another investigational drug or medical device study that has not completed primary endpoint(s) evaluation or that clinically interferes with the endpoints from this study, or subject is planning to participate in such studies prior to the completion of this study.
* Subject has had any major (e.g. cardiac, peripheral, abdominal) surgical procedure or intervention unrelated to this study within 30 days prior to the index procedure or has planned major surgical procedure or intervention within 30 days of the index procedure.
* Subject had previous bypass surgery of the target lesion.
* Subject had previously implanted stent in target lesion.
* Subject had previous treatment of the target vessel with thrombolysis or surgery.
* Subject is unwilling or unable to comply with procedures specified in the protocol or has difficulty or inability to return for follow-up visits as specified by the protocol.

Angiographic Inclusion Criteria

* The target lesion/vessel must meet all of the following angiographic criteria for the subject to participate in the trial:
* De novo lesion(s) or non-stented restenotic lesion
* Target lesion location starts at the P3 segment and terminates at 1cm above the ankle. Note: Isolated P3 lesion is not allowed. If a lesion starts in the P3 segment, it must continue into the infrapopliteal.
* Target vessel diameter ≥2 mm and ≤4 mm, based on visual estimation.
* Target lesion must have angiographic evidence of ≥70% stenosis by operator visual estimate.
* Chronic total occlusions may be included only after successful, uncomplicated wire crossing of target lesion. Successful crossing of the target lesion occurs when the tip of the guide wire is distal to the target lesion. Use of re-entry/crossing devices is not allowed. Crossing may be performed retrograde, but treatment must be performed antegrade.

Uncomplicated: Upon visual inspection, no occurrence of embolization, perforation, or occurrence of flow-limiting dissection.

* Target lesion(s) must be ≤230 mm in total lesion(s) length by operator visual estimate. A maximum of two lesions may be treated. The two lesions may be in one infrapopliteal vessel or in two distinct infrapopliteal vessels. Note: Tandem lesions may be considered a single lesion if they are separated by ≤30 mm.
* After pre-dilatation, the target lesion has ≤70% residual stenosis, absence of a flow limiting dissection (Grade D or greater) and treatable with available device matrix.
* A patent inflow artery free from significant stenosis (≥50% stenosis) as confirmed by angiography.
* At least one patent native outflow artery to the ankle or foot distal to the lesion being treated, free from significant stenosis (≥50% stenosis) as confirmed by angiography.

Angiographic Exclusion Criteria

* Aneurysm in the target vessel or proximal inflow artery.
* Inflow lesion or occlusion in the ipsilateral Iliac, SFA, popliteal arteries with length ≥15 cm.
* Significant stenosis (≥ 50%) in inflow lesion or occlusion in the ipsilateral iliac, SFA, popliteal arteries left untreated.
* Target lesion requires treatment with alternative therapy such as stenting, laser, atherectomy, cryoplasty, brachytherapy, or re-entry devices.
* Significant target vessel tortuosity or other parameters prohibiting access to the target lesion.
* Presence of thrombus in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Number of Participants with a composite of freedom from Major Adverse Limb Event (MALE) and perioperative death | 30 Days
  MALE is defined as the composite of either major amputation or major re-intervention through 30 days of the index procedure. Major amputation is defined as limb amputation above the ankle. Major re-intervention is defined as the creation of new surgical bypass graft, the use of thrombectomy or thrombolysis, or major surgical graft revision such as a jump graft or an interposition graft.
Primary Efficacy Endpoint: Rate of Late Lumen Loss (LLL) | 6 Months
  LLL is assessed by quantitative vascular angiography (QVA). LLL is the difference between minimum lumen diameter (MLD) immediately after PTA and MLD at 6 months follow-up.

SECONDARY OUTCOMES:
Rate of Device Success | Acute/Periprocedural
  Successful delivery, balloon inflation, deflation and retrieval of the intact study device
Rate of Technical Success | Acute/Periprocedural
  Successful vascular access, completion of endovascular procedure and immediate achievement of ≤ 50% residual stenosis (by core lab-assessed quantitative vascular angiography) of the treated lesion on completion of angiography.
Rate of Procedure Success | Acute/Periprocedural
  Device Success or Technical Success and the absence of procedural complications.
Rate of Restenosis | 6 Months or prior
  Assessed by Transverse-view vessel area loss percentage (TVAL%) assessed by QVA. TVAL% of the target lesion at 6 months or prior to any clinically driven target lesion revascularization (CD-TLR) of the target lesion prior to 6 months.
Number of Participants with Primary Patency | 30 Days, 6 Months, 12 Months, 24 Months
  Freedom from target vessel occlusion as determined by DUS and CD-TLR. CD-TLR is defined as any TLR of the target lesion associated with deterioration of Rutherford Class and/or increase in size of pre-existing wounds and/or occurrence of new wound(s), and lesion restenosis >50% determined by angiography.
Major Adverse Event (MAE) rate | 30 Days, 6 Months, 12 Months, 24 Months
  Composite rate of all-cause death, target limb major amputation and CD-TLR.
Amputation Free Survival | 6 Months, 12 Months, 24 Months
  Rate of subjects not requiring major amputations
Hemodynamic outcomes | 30 Days, 6 Months, 12 Months, 24 Months
  Change in ankle brachial index (ABI) and toe pressure from pre-procedure.
Change in Rutherford-Becker Classification | 30 Days, 6 Months, 12 Months, 24 Months
  Change from pre-procedure
EQ-5D | 30 Days, 6 Months, 12 Months, 24 Months
  The EQ-5D is not an abbreviation. It is a quality of Life evaluation quantified as the change from pre-procedure to time points specified below. The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'
Walking Impairment Questionnaire (WIQ) | 30 Days, 6 Months, 12 Months, 24 Months
  Walking Capacity Assessment quantified as the change from pre-procedure to time points specified below.The questions characterize patients' self-reported degree of difficulty in walking a defined distance (5, 3, 2, 1, 1/2 city blocks, 50 ft. or around the home) and speed (running/jogging one block, walking one block quickly, walking one block at average speed, or walking one block slowly). These responses are ranked on a scale of 0 to 4, (0=unable to do, 4=no difficulty). Subscale scores are determined by dividing the weighted answers by the maximum possible weighted score and multiplying by 100. Each score ranges from 0-100 with lower scores indicating lower performance. The overall score is the average of all 3 subscores.
Vascular Quality of Life Questionnaire (VascuQol) | 30 Days, 6 Months, 12 Months, 24 Months
  Quality of Life evaluation quantified as the change from pre-procedure to time points specified below. VascuQol is an instrument in which the participant is asked about their concerns, abilities, and activities. Overall values can range from 6 to 24, with a higher total sum representing better participant health.

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (3):
  - Royal Perth Hospital, Perth
  - Prince of Wales Private Hospital, Randwick
  - Royal North Shore Hospital, St Leonards
- Universitäts Klinikum Graz, Graz, Austria
- Germany (2):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - MEDINOS Kliniken des Landkreises Sonneberg GmbH, Sonneberg
- Paul Stradins University Hospital, Riga, Latvia
- Auckland City Hospital, Auckland, New Zealand